CLINICAL TRIAL: NCT04730505
Title: A Multi-center, Randomized, Pilot Trial to Evaluate the My Hematology Oncology Patient Experience (MYHOPE™) for Multiple Myeloma (MM) Digital Care Network in Patients With MM
Brief Title: A Study to Evaluate the My Hematology Oncology Patient Experience (MyHOPE™) For Multiple Myeloma (MM) Digital Care Network in Patients With MM
Acronym: MyHOPE™
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study faced multiple challenges and its launch was heavily impacted by COVID, which in turn has significantly impacted the deployment and adoption goals for a digital technology pilot. These factors led to the difficult decision to close the study.
Sponsor: Celgene (Industry)
Collaborators: Amalgam Rx (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NDS-MM-004; U1111-1263-2809 (Registry Identifier: WHO)
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Multiple Myeloma
Keywords: Digital Health; Multiple Myeloma; MYHOPE; Hematology Oncology
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient App + HCP Portal (Cohort 1) (Experimental): Cohort 1 is to assess how patients will use the Patient App if connected in real time with the Healthcare professional (HCP) Portal
  Interventions: Device: MyHOPE™ for Multiple Myeloma; Device: MyHope HCP Portal
- Patient App Alone (Cohort 2) (Experimental): Cohort 2 is to assess how patients will use the Patient App where there is no connectivity to the Healthcare professional (HCP) Portal and thus no real-time data sharing with the HCP Portal
  Interventions: Device: MyHOPE™ for Multiple Myeloma

INTERVENTIONS:
Device: MyHOPE™ for Multiple Myeloma — The MyHOPE for MM Platform is designed to provide patients with tools and resources to support them in their overall experience with MM. Patients can share their data through a PDF or by showing their device to their care team at clinic visits.
Device: MyHope HCP Portal — Is designed to provide HCPs with the ability to view patient data and symptom notifications (Cohort 1 only) to provide support between clinic visits and to facilitate dialogue during clinic visits.
  Arms: Patient App + HCP Portal (Cohort 1)

SUMMARY:
NDS-MM-004 is a multi-center, randomized, pilot trial to evaluate the MyHOPE for multiple myeloma (MM) Platform in patients with MM. The MyHOPE for MM Platform is a validated investigational device manufactured by Amalgam Rx, Inc. and designed to provide patients with a comprehensive set of tools and resources to support the patient throughout their overall experience with MM.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old with a diagnosis of Multiple Myeloma
* Patient must reside in the USA.
* Patients within each of the following subgroups, at one of the following timepoints, will be eligible for entry:

  1. Newly-diagnosed multiple myeloma transplant-eligible
  2. Patients undergoing their first ASCT
  3. Newly-diagnosed multiple myeloma transplant-ineligible
  4. Relapsed and/or refractory.

Exclusion Criteria:

* Patient has a condition(s) that, in the opinion of the Investigator, would make participation infeasible such as inability to provide informed consent, illiteracy, or inability to speak, read, and write in English.
* Patient is on hospice.
* Patient is receiving or has received an investigational agent < 28 days prior to randomization or during this pilot study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Monthly eligibility and recruitment rates per month of patients with multiple myeloma | Up to 12 months
  is defined as the number of patients with MM that satisfied entry criteria per study site/month)
User average weekly log-in rates over the duration of follow-up from patients with MM and HCPs | Up to 6 months
  is defined as the number of times a user attempts to log in/week
Duration of follow-up | Up to 6 months
  is defined as the mean, median, and range of time from each user's first login to his or her last login to the Patient App or to the HCP Portal
Patient-reported outcome completion rates | Up to 6 months
  Is defined as the number of data points that are completed divided by the number of data points that could have been completed at each specified timepoint, relative to the enrollment date of each participant
Frequency of user access by feature and by month, relative to the enrollment date of each participant | Up to 6 months
  Is defined as how often patients access various features of the app, per month relative to the enrollment date of each participant
Percentage of patients for whom the HCPs complete the 6-month assessments | up to 18 months
  is defined as number of patients for whom HCPs provided 6-month assessments [eg, disease response assessments] divided by the number of patients for whom HCPs provided baseline data)
Patient empowerment and self-efficacy measured by CASE-Cancer | Up to 6 months
  The instrument consists of 3 subscales: understanding and participating in care, maintaining a positive attitude, and seeking and obtaining information. All items are scored on a range of 1 to 4 from strongly disagree to strongly agree, with higher score indicating better empowerment

SECONDARY OUTCOMES:
Proportion of respondents scoring 4 or 5 on the Patient Platform Usability Survey or Healthcare Provider Platform Survey | Up to 18 months
  is defined as the number of respondents giving a score of 4 or 5 to each of the questions in the Patient Platform Usability Survey divided by overall number of respondents for that question or number of respondents giving a score of 4 or 5 to each of the questions in the Healthcare Provider Platform Usability Survey divided by overall number of respondents for that question, respectively
Quality of life measured by Functional Assessment of Cancer Therapy-Multiple Myeloma (FACT-MM) total score | Up to 6 months
  This scale addresses symptoms and functional limitations that are important to patients with MM. The items are scored on a 0 ("Not at all") to 4 ("Very much") response scale.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ludwig, Study Director — Bristol-Myers Squibb
Locations (34):
- United States (34):
  - Mitchell Cancer Center, University of South Alabama, Mobile, Alabama
  - Mayo Cliinic - Scottsdale, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - James R Berenson MD Inc, West Hollywood, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Cancer Specialists of North Florida - Jacksonville, Jacksonville, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Augusta University - Georgia Cancer Center, Augusta, Georgia
  - Innovation Clinical Research of the Pacific, Honolulu, Hawaii
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - American Oncology Partner Maryland, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Western Michigan Cancer Center, Kalamazoo, Michigan
  - Newland Medical Associates, PC, Southfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NY Cancer and Blood Specialists, Port Jefferson Station, New York
  - Rochester General Hospital - Lipson Cancer Institute, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Tri County Hematology Oncology, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Jefferson Medical Oncology Associates, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - West Cancer Center, Germantown, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Community Cancer Trials of Utah, Ogden, Utah

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/